CLINICAL TRIAL: NCT00882960
Title: Atomization of Fentanyl: A Randomized Comparison Study of Intranasal Versus Intravenous Fentanyl for Pre-hospital Pain Management
Brief Title: Intranasal Fentanyl for Pain Management
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genesys (Other)
Responsible Party: Dr. Ryan Kirby, M.D., Genesys Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104904-1
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Trauma; Pain
Keywords: pre-hospital; intra-nasal fentanyl; patients requiring analgesia
MeSH Terms: conditions — Wounds and Injuries; Pain

ARMS (2):
- 1 (Active Comparator): patients who are randomized to receive intravenous fentanyl for control of their pain
  Interventions: Drug: intravenous fentanyl
- 2 (Active Comparator): patients who are randomized to receive intra-nasal fentanyl for control of their pain
  Interventions: Drug: intra-nasal fentanyl

INTERVENTIONS:
Drug: intravenous fentanyl — An IV will be established and used to deliver Fentanyl at 50 micrograms to patients who meet pre-hospital protocol for pain management. Examples of this may be burn patients, fractures, trauma.
  Arms: 1
Drug: intra-nasal fentanyl — a mucosal atomization device will be used to deliver 50 mcg of Fentanyl to patients who have been identified at requiring pre-hospital pain management
  Arms: 2

SUMMARY:
Goal of the research will be to demonstrate a reduction in reported pain following the atomization and intra-nasal administration of Fentanyl versus the reduction in pain achieved from intravenous Fentanyl. It is hypothesized that pain should be reduced following fentanyl administration using the intra-nasal atomization equal to the intravenous delivery.

DETAILED DESCRIPTION:
Currently, pre-hospital providers have the ability to administer analgesia to patients through only intravenous routes. Often times patients have been exposed to the elements, present with poor anatomy, or are in such a position that makes establishing intravenous impractical or impossible. The lack of delivery method than prevents the patients from receiving humane and indicated pain medication. In patients who access is achieved, they are first subjected to a painful procedure that often will be repeated within twenty-four hours by most hospital policies and than subjects them to potential infection risk, being often times in less than aseptic conditions.

The goal of the study will be to test the method of administration of pain medication using atomization through an intra-nasal route as compared to the current standard of drug administration intravenous. The medication to be administered will be Fentanyl, a previously established and approved pre-hospital analgesic medication. As with any drug there are potential risks associated with unknown side effects or allergies, the risk would not be enhanced given the use of a different delivery device. Specific risks associated with the use of this delivery route would include but not be limited to potential soft tissue injuries, epistaxis, and aspiration

The study will measure reduction in pain following the delivery of atomized fentanyl via intra-nasal administration as compared with intravenous. We will ask participants to quantify their pain using the Wong-Baker FACES pain scale (previously established valid instrument of pain assessment) and assign a number to the pain they are feeling. The drug will than be administered using the atomizer and two subsequent reports of pain using the same scale will be taken along with vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Persons who meet the current State of Michigan County of Oakland and County of Genesee pre-hospital pain requiring analgesia.
* Examples of these patients would be those with fractures, kidney stones, or traumatic injuries, burns.

Exclusion Criteria:

* Patients who have compromised nasal pharynx such as those who have obvious fractures or epistaxis.
* Additionally patients who are in the supine position for cervical spine immobilization will be excluded.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The primary measure will be the change recorded in patients subjective pain using a standardized scale | Pain will be assessed at 5 and 10 minutes post administration of Fentanyl

SECONDARY OUTCOMES:
Change in patients vital signs: blood pressure, respiratory rate, heart rate, pulse oximetry will be monitored at 5 and 10 minutes following Atomized Fentanyl | 5 and 10 minutes post medication delivery

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Janssen, D.O., Study Chair — Director of Emergency Medicine Residency, Genesys Regional Medical Center; Ryan P Kirby, M.D., Principal Investigator — Resident physician, Genesys Regional Medical Center; Stuart Etengoff, D.O., Study Director — Core Faculty, Department of Emergency Medicine, Genesys Regional Medical Center
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States